CLINICAL TRIAL: NCT04966780
Title: Dose-response Relation Between the Development of a Refeeding-like Syndrome and Sodium Balance in Patients Undergoing Acute Abdominal Surgery
Brief Title: Refeeding Like Syndrome in Acute Disease
Acronym: RLS
Status: Completed | Type: Observational
Sponsor: Jens Rikardt Andersen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Associate Professor, Primary Investigator, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: RLS in surgery
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Refeeding Syndrome; Acute Abdomen
Keywords: refeeding syndrome; acute abdominal disease
MeSH Terms: conditions — Refeeding Syndrome; Abdomen, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: acute abdominal surgery — Acute surgery for acute abdominal disease

SUMMARY:
The refeeding syndrome has been reported without any evidence of prolopnged semistarvation, thus being different from the traditional disease.

The investigators wanted to investigate, if sodium infusions could be part of the explanation.

DETAILED DESCRIPTION:
Background: Refeeding syndrome is conventionally connected to start of feeding after prolonged periods of semi-starvation and adaption. However, it is also described in acutely ill patients and in ICU patients without a history of adaption, but sometimes only defined as a drop in p-phosphate without clinical manifestations. The investigators hypothesize, that a positive sodium balance could induce the refeeding-like syndrome (RLS).

Method: Consecutive patients for acute, abdominal surgery were included and observed until discharge or up to seven days postoperatively with daily sodium and phosphate balance measurements.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 yr
* ready for acute surgery
* able to understand and cooperate.

Exclusion Criteria:

* pregnancy or breastfeeding
* renal insufficiency (p-creatinine>400 micr mol/l)
* re-operations
* expected hospital stay < 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive, adult patients for acute, abdominal surgery were asked top be included and observed until discharge or up to seven days postoperatively with daily sodium and phosphate balance measurements.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
sodium balance | 7 days
  correlation between sodium balance and occurrence of the refeeding syndrome

SECONDARY OUTCOMES:
plasma phosphate | 7 days
  correlation between sodium balance and change in plasma phosphate
urinary excretion of phosphate | 7 days
  correletion between sodium balance and urinary excretion of phosphate
phosphate balance | 7 days
  correlation between decline in plasma phosphate and urinary excretion of phosphate

CONTACTS AND LOCATIONS:
Overall Officials: jens R Andersen, Principal Investigator — University of Copenhagen
Locations (1):
- Herlev University Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No